CLINICAL TRIAL: NCT04009499
Title: A Multicenter, Open-Label Extension Study to Assess the Long-Term Safety, Tolerability, and Efficacy of Bimekizumab in the Treatment of Subjects With Active Psoriatic Arthritis
Brief Title: A Study to Assess the Long-term Safety, Tolerability, and Efficacy of Bimekizumab in the Treatment of Subjects With Active Psoriatic Arthritis
Acronym: BE VITAL
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PA0012; 2018-004725-86 (EudraCT Number); 2023-506528-95 (Registry Identifier: EU Clinical Trials); U1111-1304-6874 (Other: World Health Organization (WHO))
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic Arthritis; PsA; Bimekizumab
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — bimekizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bimekzumab dosage regimen (Experimental): Subjects participating in the study will receive assigned bimekizumab dosage regimen during the Treatment Period.
  Interventions: Drug: Bimekizumab

INTERVENTIONS:
Drug: Bimekizumab — Subjects will receive bimekizumab at pre-specified time-points.
  Other Names: BKZ; UCB4940

SUMMARY:
This is a study to assess the long-term safety, long-term efficacy and tolerability of bimekizumab administered subcutaneously (sc) in adult subjects with psoriatic arthritis (PsA).

ELIGIBILITY:
Inclusion Criteria:

* In the opinion of the Investigator, the subject is expected to benefit from participation in this Open-Label Extension study
* Subject completed PA0010 [NCT03895203] or PA0011 [NCT03896581] without meeting any withdrawal criteria
* Female subjects must be postmenopausal, permanently sterilized or willing to use a highly effective method of contraception

Exclusion Criteria:

* Female subjects who plan to become pregnant during the study or within 20 weeks following the last dose of investigational medicinal product (IMP)
* Subjects who meet any withdrawal criteria in PA0010 or PA0011. For any subject with an ongoing serious adverse event (SAE), or a history of serious infections (including hospitalizations) in the feeder studies, the Medical Monitor must be consulted prior to the subject's entry into PA0012, although the decision to enroll the subject remains with the Investigator
* Subject has a positive or 2 indeterminate interferon gamma release assays (IGRAs) in one of the feeder studies, unless appropriately evaluated and treated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1131 (Actual)
Dates: Start 2019-08-13 (Actual); Primary Completion 2026-05-25 (Estimated); Study Completion 2026-05-25 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) during the study | From PA0012 Entry Visit until Safety Follow-Up (up to Week 212)
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Incidence of treatment-emergent serious adverse events (SAEs) during the study | From PA0012 Entry Visit until Safety Follow-Up (up to Week 212)
  A serious adverse event (SAE) is any untoward medical occurrence that at any dose:
  * Results in death
  * Is life-threatening
  * Requires in patient hospitalization or prolongation of existing hospitalization
  * Is a congenital anomaly or birth defect
  * Is an infection that requires treatment parenteral antibiotics
  * Other important medical events which based on medical or scientific judgement may jeopardize the patients, or may require medical or surgical intervention to prevent any of the above

SECONDARY OUTCOMES:
TEAEs leading to withdrawal from investigational medicinal product (IMP) during the study | From PA0012 Entry Visit until Safety Follow-Up (up to Week 212)
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
American College of Rheumatology 20% improvement (ACR20) response at Week 24 in PA0012 using the Baseline of PA0010 or PA0011 | Baseline of PA0010 or PA0011, Week 24 in PA0012
  The ACR20 response rate is based on a 20% or greater improvement of arthritis relative to Baseline of PA0010 or PA0011.
American College of Rheumatology 20% improvement (ACR20) response at Week 52 in PA0012 using the Baseline of PA0010 or PA0011 | Baseline of PA0010 or PA0011, Week 52 in PA0012
  The ACR20 response rate is based on a 20% or greater improvement of arthritis relative to Baseline of PA0010 or PA0011.
American College of Rheumatology 20% improvement (ACR20) response at Week 140 in PA0012 using the Baseline of PA0010 or PA0011 | Baseline of PA0010 or PA0011, Week 140 in PA0012
  The ACR20 response rate is based on a 20% or greater improvement of arthritis relative to Baseline of PA0010 or PA0011.
American College of Rheumatology 50% improvement (ACR50) response at Week 24 in PA0012 using the Baseline of PA0010 or PA0011 | Baseline of PA0010 or PA0011, Week 24 in PA0012
  The ACR50 response rate is based on a 50% or greater improvement of arthritis relative to Baseline of PA0010 or PA0011.
American College of Rheumatology 50% improvement (ACR50) response at Week 52 in PA0012 using the Baseline of PA0010 or PA0011 | Baseline of PA0010 or PA0011, Week 52 in PA0012
  The ACR50 response rate is based on a 50% or greater improvement of arthritis relative to Baseline of PA0010 or PA0011.
American College of Rheumatology 50% improvement (ACR50) response at Week 140 in PA0012 using the Baseline of PA0010 or PA0011 | Baseline of PA0010 or PA0011, Week 140 in PA0012
  The ACR50 response rate is based on a 50% or greater improvement of arthritis relative to Baseline of PA0010 or PA0011.
American College of Rheumatology 70% improvement (ACR70) response at Week 24 in PA0012 using the Baseline of PA0010 or PA0011 | Baseline of PA0010 or PA0011, Week 24 in PA0012
  The ACR70 response rate is based on a 70% or greater improvement of arthritis relative to Baseline of PA0010 or PA0011.
American College of Rheumatology 70% improvement (ACR70) response at Week 52 in PA0012 using the Baseline of PA0010 or PA0011 | Baseline of PA0010 or PA0011, Week 52 in PA0012
  The ACR70 response rate is based on a 70% or greater improvement of arthritis relative to Baseline of PA0010 or PA0011.
American College of Rheumatology 70% improvement (ACR70) response at Week 140 in PA0012 using the Baseline of PA0010 or PA0011 | Baseline of PA0010 or PA0011, Week 140 in PA0012
  The ACR70 response rate is based on a 70% or greater improvement of arthritis relative to Baseline of PA0010 or PA0011.
Psoriasis Area Severity Index 75 (PASI75) response at Week 24 in PA0012 using the Baseline of PA0010 or PA0011 | Baseline of PA0010 or PA0011, Week 24 in PA0012
  The PASI will be assessed for the purposes of determining response only in subjects with psoriasis (PSO) involving at ≥3% of body surface area (BSA) at Baseline of PA0010 or PA0011.
  The PASI75 response is based on at least 75% improvement in the PASI score compared to Baseline of of PA0010 or PA0011.
  The Investigator assesses the average redness, thickness, and scaliness of lesions in each body area (each on a 5-point scale); 0=none, 1=slight, 2=moderate, 3=marked, and 4=very marked. The PASI score ranges from 0 to 72 with a higher score indicating increased disease severity.
Psoriasis Area Severity Index 75 (PASI75) response at Week 52 in PA0012 using the Baseline of PA0010 or PA0011 | Baseline of PA0010 or PA0011, Week 52 in PA0012
  The PASI will be assessed for the purposes of determining response only in subjects with psoriasis (PSO) involving at ≥3% of body surface area (BSA) at Baseline of PA0010 or PA0011.
  The PASI75 response is based on at least 75% improvement in the PASI score compared to Baseline of of PA0010 or PA0011.
  The Investigator assesses the average redness, thickness, and scaliness of lesions in each body area (each on a 5-point scale); 0=none, 1=slight, 2=moderate, 3=marked, and 4=very marked. The PASI score ranges from 0 to 72 with a higher score indicating increased disease severity.
Psoriasis Area Severity Index 75 (PASI75) response at Week 140 in PA0012 using the Baseline of PA0010 or PA0011 | Baseline of PA0010 or PA0011, Week 140 in PA0012
  The PASI will be assessed for the purposes of determining response only in subjects with psoriasis (PSO) involving at ≥3% of body surface area (BSA) at Baseline of PA0010 or PA0011.
  The PASI75 response is based on at least 75% improvement in the PASI score compared to Baseline of of PA0010 or PA0011.
  The Investigator assesses the average redness, thickness, and scaliness of lesions in each body area (each on a 5-point scale); 0=none, 1=slight, 2=moderate, 3=marked, and 4=very marked. The PASI score ranges from 0 to 72 with a higher score indicating increased disease severity.
Psoriasis Area Severity Index 90 (PASI90) response at Week 24 in PA0012 using the Baseline of PA0010 or PA0011 | Baseline of PA0010 or PA0011, Week 24 in PA0012
  The PASI will be assessed for the purposes of determining response only in subjects with psoriasis (PSO) involving at ≥3% of body surface area (BSA) at Baseline of PA0010 or PA0011.
  The PASI90 response is based on at least 90% improvement in the PASI score compared to Baseline of of PA0010 or PA0011.
  The Investigator assesses the average redness, thickness, and scaliness of lesions in each body area (each on a 5-point scale); 0=none, 1=slight, 2=moderate, 3=marked, and 4=very marked. The PASI score ranges from 0 to 72 with a higher score indicating increased disease severity.
Psoriasis Area Severity Index 90 (PASI90) response at Week 52 in PA0012 using the Baseline of PA0010 or PA0011 | Baseline of PA0010 or PA0011, Week 52 in PA0012
  The PASI will be assessed for the purposes of determining response only in subjects with psoriasis (PSO) involving at ≥3% of body surface area (BSA) at Baseline of PA0010 or PA0011.
  The PASI90 response is based on at least 90% improvement in the PASI score compared to Baseline of of PA0010 or PA0011.
  The Investigator assesses the average redness, thickness, and scaliness of lesions in each body area (each on a 5-point scale); 0=none, 1=slight, 2=moderate, 3=marked, and 4=very marked. The PASI score ranges from 0 to 72 with a higher score indicating increased disease severity.
Psoriasis Area Severity Index 90 (PASI90) response at Week 140 in PA0012 using the Baseline of PA0010 or PA0011 | Baseline of PA0010 or PA0011, Week 140 in PA0012
  The PASI will be assessed for the purposes of determining response only in subjects with psoriasis (PSO) involving at ≥3% of body surface area (BSA) at Baseline of PA0010 or PA0011.
  The PASI90 response is based on at least 90% improvement in the PASI score compared to Baseline of of PA0010 or PA0011.
  The Investigator assesses the average redness, thickness, and scaliness of lesions in each body area (each on a 5-point scale); 0=none, 1=slight, 2=moderate, 3=marked, and 4=very marked. The PASI score ranges from 0 to 72 with a higher score indicating increased disease severity.
Investigator Global Assessment (IGA) score of 0 (clear) or 1 (almost clear) AND at least a 2-grade reduction at Week 24 from the Baseline of PA0010 or PA0011 | Baseline of PA0010 or PA0011, Week 24 in PA0012
  A static Investigator Global Assessment (IGA) for psoriasis (PSO) will be used to assess disease severity during the study only for subjects with IGA ≥2 at the Baseline of PA0010 or PA0011.
  An IGA response is defined as Clear or Almost Clear with at least a 2-category improvement relative to Baseline of PA0010 or PA0011.
Investigator Global Assessment (IGA) score of 0 (clear) or 1 (almost clear) AND at least a 2-grade reduction at Week 52 from the Baseline of PA0010 or PA0011 | Baseline of PA0010 or PA0011, Week 52 in PA0012
  A static Investigator Global Assessment (IGA) for psoriasis (PSO) will be used to assess disease severity during the study only for subjects with IGA ≥2 at the Baseline of PA0010 or PA0011.
  An IGA response is defined as Clear or Almost Clear with at least a 2-category improvement relative to Baseline of PA0010 or PA0011.
Investigator Global Assessment (IGA) score of 0 (clear) or 1 (almost clear) AND at least a 2-grade reduction at Week 140 from the Baseline of PA0010 or PA0011 | Baseline of PA0010 or PA0011, Week 140 in PA0012
  A static Investigator Global Assessment (IGA) for psoriasis (PSO) will be used to assess disease severity during the study only for subjects with IGA ≥2 at the Baseline of PA0010 or PA0011.
  An IGA response is defined as Clear or Almost Clear with at least a 2-category improvement relative to Baseline of PA0010 or PA0011
Enthesitis-free state based on the Leeds Enthesitis Index (LEI) at Week 24 in PA0012 using the subgroup of subjects with enthesitis at the Baseline of PA0010 or PA0011 | Baseline of PA0010 or PA0011, Week 24 in PA0012
  Presence of enthesitis will be assessed in the subgroup of subjects with enthesitis by palpation on the lateral epicondyles of the humerus (elbows), medial femoral epicondyles (knees), and Achilles tendons (heels) bilaterally and scored as 0=no pain and 1=painful at Baseline of PA0010 or PA0011.
Enthesitis-free state based on the Leeds Enthesitis Index (LEI) at Week 52 in PA0012 using the subgroup of subjects with enthesitis at the Baseline of PA0010 or PA0011 | Baseline of PA0010 or PA0011, Week 52 in PA0012
  Presence of enthesitis will be assessed in the subgroup of subjects with enthesitis by palpation on the lateral epicondyles of the humerus (elbows), medial femoral epicondyles (knees), and Achilles tendons (heels) bilaterally and scored as 0=no pain and 1=painful at Baseline of PA0010 or PA0011.
Enthesitis-free state based on the Leeds Enthesitis Index (LEI) at Week 140 in PA0012 using the subgroup of subjects with enthesitis at the Baseline of PA0010 or PA0011 | Baseline of PA0010 or PA0011, Week 140 in PA0012
  Presence of enthesitis will be assessed in the subgroup of subjects with enthesitis by palpation on the lateral epicondyles of the humerus (elbows), medial femoral epicondyles (knees), and Achilles tendons (heels) bilaterally and scored as 0=no pain and 1=painful at Baseline of PA0010 or PA0011.
Enthesitis-free state based on the Spondyloarthritis Research Consortium of Canada (SPARCC) index at Week 24 in PA0012 using the subgroup of subjects with enthesitis at the Baseline of PA0010 or PA0011 | Baseline of PA0010 or PA0011, Week 24 in PA0012
  Presence of enthesitis will be assessed in the subgroup of subjects with enthesitis at Baseline of PA0010 or PA0011. The Spondyloarthritis Research Consortium of Canada (SPARCC) is an index that measures the severity of enthesitis through the assessment of 16 sites. Tenderness on examination is recorded as either present (1) or absent (0) for each of the 16 sites, for an overall score range of 0 to 16.
Enthesitis-free state based on the Spondyloarthritis Research Consortium of Canada (SPARCC) index at Week 52 in PA0012 using the subgroup of subjects with enthesitis at the Baseline of PA0010 or PA0011 | Baseline of PA0010 or PA0011, Week 52 in PA0012
  Presence of enthesitis will be assessed in the subgroup of subjects with enthesitis at Baseline of PA0010 or PA0011. The Spondyloarthritis Research Consortium of Canada (SPARCC) is an index that measures the severity of enthesitis through the assessment of 16 sites. Tenderness on examination is recorded as either present (1) or absent (0) for each of the 16 sites, for an overall score range of 0 to 16.
Enthesitis-free state based on the Spondyloarthritis Research Consortium of Canada (SPARCC) index at Week 140 in PA0012 using the subgroup of subjects with enthesitis at the Baseline of PA0010 or PA0011 | Baseline of PA0010 or PA0011, Week 140 in PA0012
  Presence of enthesitis will be assessed in the subgroup of subjects with enthesitis at Baseline of PA0010 or PA0011. The Spondyloarthritis Research Consortium of Canada (SPARCC) is an index that measures the severity of enthesitis through the assessment of 16 sites. Tenderness on examination is recorded as either present (1) or absent (0) for each of the 16 sites, for an overall score range of 0 to 16.
Dactylitis-free state based on the Leeds Dactylitis Index (LDI) at Week 24 in PA0012 using the subgroup of subjects with dactylitis at the Baseline of PA0010 or PA0011 | Baseline of PA0010 or PA0011, Week 24 in PA0012
  Presence of dactylitis will be assessed in the subgroup of subjects with dactylitis using the LDI basic which evaluates for a >=10% difference in the circumference of the digit compared to the opposite digit this is then multiplied by the tenderness score, using a simple grading system (0=absent, 1=present) at Baseline of PA0010 or PA0011.
Dactylitis-free state based on the Leeds Dactylitis Index (LDI) at Week 52 in PA0012 using the subgroup of subjects with dactylitis at the Baseline of PA0010 or PA0011 | Baseline of PA0010 or PA0011, Week 52 in PA0012
  Presence of dactylitis will be assessed in the subgroup of subjects with dactylitis using the LDI basic which evaluates for a >=10% difference in the circumference of the digit compared to the opposite digit this is then multiplied by the tenderness score, using a simple grading system (0=absent, 1=present) at Baseline of PA0010 or PA0011.
Dactylitis-free state based on the Leeds Dactylitis Index (LDI) at Week 140 in PA0012 using the subgroup of subjects with dactylitis at the Baseline of PA0010 or PA0011 | Baseline of PA0010 or PA0011, Week 140 in PA0012
  Presence of dactylitis will be assessed in the subgroup of subjects with dactylitis using the LDI basic which evaluates for a >=10% difference in the circumference of the digit compared to the opposite digit this is then multiplied by the tenderness score, using a simple grading system (0=absent, 1=present) at Baseline of PA0010 or PA0011.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (138):
- United States (31):
  - Pa0012 50017, Phoenix, Arizona
  - Pa0012 50035, San Diego, California
  - Pa0012 50033, Palm Harbor, Florida
  - Pa0012 50037, Tampa, Florida
  - Pa0012 50039, Atlanta, Georgia
  - Pa0012 50024, Boise, Idaho
  - Pa0012 50028, Lexington, Kentucky
  - Pa0012 50023, Baton Rouge, Louisiana
  - Pa0012 50015, Hagerstown, Maryland
  - Pa0012 50047, Boston, Massachusetts
  - Pa0012 50019, Lansing, Michigan
  - Pa0012 50016, St Louis, Missouri
  - Pa0012 50005, Freehold, New Jersey
  - Pa0012 50029, Albuquerque, New Mexico
  - Pa0012 50010, Brooklyn, New York
  - Pa0012 50011, New York, New York
  - Pa0012 50034, Rochester, New York
  - Pa0012 50125, Charlotte, North Carolina
  - Pa0012 50031, Salisbury, North Carolina
  - Pa0012 50040, Vandalia, Ohio
  - Pa0012 50020, Duncansville, Pennsylvania
  - Pa0012 50006, Wyomissing, Pennsylvania
  - Pa0012 50008, Johnston, Rhode Island
  - Pa0012 50007, Orangeburg, South Carolina
  - Pa0012 50001, Jackson, Tennessee
  - Pa0012 50012, Memphis, Tennessee
  - Pa0012 50002, Austin, Texas
  - Pa0012 50049, Corpus Christi, Texas
  - Pa0012 50036, Mesquite, Texas
  - Pa0012 50009, Waco, Texas
  - Pa0012 50050, Beckley, West Virginia
- Australia (6):
  - Pa0012 30005, Camberwell
  - Pa0012 30002, Clayton
  - Pa0012 30008, Hobart
  - Pa0012 30003, Maroochydore
  - Pa0012 30007, Victoria Park
  - Pa0012 30006, Woodville South
- Belgium (3):
  - Pa0012 40003, Genk
  - Pa0012 40002, Leuven
  - Pa0012 40059, Mons
- Canada (4):
  - Pa0012 50041, Québec
  - Pa0012 50042, Rimouski
  - Pa0012 50043, Sydney
  - Pa0012 50044, Trois-Rivières
- Czechia (11):
  - Pa0012 40061, Brno
  - Pa0012 40065, Brno
  - Pa0012 40062, Moravska Ostrava A Privoz
  - Pa0012 40009, Pardubice
  - Pa0012 40013, Prague
  - Pa0012 40014, Prague
  - Pa0012 40015, Prague
  - Pa0012 40063, Prague
  - Pa0012 40066, Prague
  - Pa0012 40010, Uherské Hradiště
  - Pa0012 40012, Zlín
- France (2):
  - Pa0012 40068, Chambray-lès-Tours
  - Pa0012 40019, Paris
- Germany (10):
  - Pa0012 40074, Bad Doberan
  - Pa0012 40025, Berlin
  - Pa0012 40076, Cottbus
  - Pa0012 40023, Erlangen
  - Pa0012 40117, Frankfurt am Main
  - Pa0012 40029, Hamburg
  - Pa0012 40071, Hamburg
  - Pa0012 40027, Herne
  - Pa0012 40078, Leipzig
  - Pa0012 40026, Ratingen
- Hungary (7):
  - Pa0012 40081, Budapest
  - Pa0012 40083, Budapest
  - Pa0012 40032, Debrecen
  - Pa0012 40030, Eger
  - Pa0012 40082, Kistarcsa
  - Pa0012 40079, Szentes
  - Pa0012 40033, Székesfehérvár
- Italy (3):
  - Pa0012 40084, Catania
  - Pa0012 40087, Milan
  - Pa0012 40086, Reggio Emilia
- Japan (14):
  - Pa0012 20035, Bunkyō City
  - Pa0012 20030, Chūōku
  - Pa0012 20043, Itabashi-ku
  - Pa0012 20036, Kawachi-Nagano
  - Pa0012 20045, Kita-gun
  - Pa0012 20049, Kitakyushu
  - Pa0012 20044, Minatoku
  - Pa0012 20033, Nagoya
  - Pa0012 20041, Osaka
  - Pa0012 20046, Osaka
  - Pa0012 20048, Saitama
  - Pa0012 20031, Sapporo
  - Pa0012 20042, Sasebo
  - Pa0012 20032, Suita
- Poland (19):
  - Pa0012 40093, Bialystok
  - Pa0012 40119, Bydgoszcz
  - Pa0012 40038, Elblag
  - Pa0012 40088, Elblag
  - Pa0012 40096, Gdynia
  - Pa0012 40042, Krakow
  - Pa0012 40092, Krakow
  - Pa0012 40037, Lublin
  - Pa0012 40091, Nowa Sól
  - Pa0012 40044, Poznan
  - Pa0012 40090, Poznan
  - Pa0012 40041, Warsaw
  - Pa0012 40094, Warsaw
  - Pa0012 40097, Warsaw
  - Pa0012 40098, Warsaw
  - Pa0012 40118, Warsaw
  - Pa0012 40039, Wroclaw
  - Pa0012 40043, Wroclaw
  - Pa0012 40095, Wroclaw
- Russia (17):
  - Pa0012 20002, Moscow
  - Pa0012 20005, Moscow
  - Pa0012 20010, Moscow
  - Pa0012 20017, Moscow
  - Pa0012 20013, Petrozavodsk
  - Pa0012 20012, Ryazan
  - Pa0012 20016, Ryazan
  - Pa0012 20001, Saint Petersburg
  - Pa0012 20003, Saint Petersburg
  - Pa0012 20004, Saint Petersburg
  - Pa0012 20009, Saint Petersburg
  - Pa0012 20083, Saint Petersburg
  - Pa0012 20007, Saratov
  - Pa0012 20014, Ulyanovsk
  - Pa0012 20006, Vladimir
  - Pa0012 20008, Yaroslavl
  - Pa0012 20015, Yaroslavl
- Spain (8):
  - Pa0012 40045, A Coruña
  - Pa0012 40105, Córdoba
  - Pa0012 40102, Málaga
  - Pa0012 40101, Sabadell
  - Pa0012 40104, Santiago de Compostela
  - Pa0012 40049, Seville
  - Pa0012 40106, Seville
  - Pa0012 40099, Vigo
- United Kingdom (3):
  - Pa0012 40109, Oxford
  - Pa0012 40116, Peterborough
  - Pa0012 40107, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this study may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: http://www.Vivli.org

REFERENCES:
- [Result] Mease PJ, Warren RB, Nash P, Grouin JM, Lyris N, Willems D, Taieb V, Eells J, McInnes IB. Comparative Effectiveness of Bimekizumab and Risankizumab in Patients with Psoriatic Arthritis at 52 Weeks Assessed Using a Matching-Adjusted Indirect Comparison. Rheumatol Ther. 2024 Oct;11(5):1403-1412. doi: 10.1007/s40744-024-00706-w. Epub 2024 Aug 9. PMID 39120849
- [Result] Gossec L, Orbai AM, de Wit M, Coates LC, Ogdie A, Ink B, Coarse J, Lambert J, Taieb V, Gladman DD. Effect of bimekizumab on patient-reported disease impact in patients with psoriatic arthritis: 1-year results from two phase 3 studies. Rheumatology (Oxford). 2024 Sep 1;63(9):2399-2410. doi: 10.1093/rheumatology/keae277. PMID 38754125
- [Result] Kristensen LE, Tillett W, Nash P, Coates LC, Mease PJ, Ogdie A, Gisondi P, Ink B, Prickett AR, Bajracharya R, Taieb V, Lyris N, Lambert J, Walsh JA. Association of achieving clinical disease control criteria and patient-reported outcomes in bimekizumab-treated patients with active psoriatic arthritis: results from two phase III studies. Ther Adv Musculoskelet Dis. 2024 Nov 11;16:1759720X241288071. doi: 10.1177/1759720X241288071. eCollection 2024. PMID 39534481
- [Result] Mease PJ, Merola JF, Tanaka Y, Gossec L, McInnes IB, Ritchlin CT, Landewe RBM, Asahina A, Ink B, Heinrichs A, Bajracharya R, Shende V, Coarse J, Coates LC. Summary of Research: Safety and Efficacy of Bimekizumab in Patients with Psoriatic Arthritis: 2-Year Results from Two Phase 3 Studies. Rheumatol Ther. 2025 Aug;12(4):609-612. doi: 10.1007/s40744-025-00764-8. Epub 2025 May 10. PMID 40347389
- [Result] Thaci D, Asahina A, Boehncke WH, Gottlieb AB, Lebwohl M, Warren RB, Edens H, Ink B, Bajracharya R, Coarse J, Merola JF. Bimekizumab Efficacy and Safety in Patients with Psoriatic Arthritis with Substantial Skin and Nail Psoriasis to 1 Year. Dermatol Ther (Heidelb). 2025 Dec 12. doi: 10.1007/s13555-025-01599-5. Online ahead of print. PMID 41381988
- [Derived] Mease PJ, Gensler LS, Orbai AM, Warren RB, Bajracharya R, Ink B, Marten A, Massow U, Shende V, Manente M, Peterson L, White K, Landewe R, Poddubnyy D. Long-term safety of bimekizumab in adult patients with axial spondyloarthritis or psoriatic arthritis: pooled results from integrated phase IIb/III clinical studies. RMD Open. 2025 Apr 6;11(2):e005026. doi: 10.1136/rmdopen-2024-005026. PMID 40194794
- [Derived] Mease PJ, Merola JF, Tanaka Y, Gossec L, McInnes IB, Ritchlin CT, Landewe RBM, Asahina A, Ink B, Heinrichs A, Bajracharya R, Shende V, Coarse J, Coates LC. Safety and Efficacy of Bimekizumab in Patients with Psoriatic Arthritis: 2-Year Results from Two Phase 3 Studies. Rheumatol Ther. 2024 Oct;11(5):1363-1382. doi: 10.1007/s40744-024-00708-8. Epub 2024 Aug 31. PMID 39215949
- [Derived] Warren RB, McInnes IB, Nash P, Grouin JM, Lyris N, Willems D, Taieb V, Eells J, Mease PJ. Comparative Effectiveness of Bimekizumab and Guselkumab in Patients with Psoriatic Arthritis at 52 Weeks Assessed Using a Matching-Adjusted Indirect Comparison. Rheumatol Ther. 2024 Jun;11(3):829-839. doi: 10.1007/s40744-024-00659-0. Epub 2024 Mar 15. PMID 38488975
- [Derived] Mease PJ, Warren RB, Nash P, Grouin JM, Lyris N, Willems D, Taieb V, Eells J, McInnes IB. Comparative Effectiveness of Bimekizumab and Secukinumab in Patients with Psoriatic Arthritis at 52 Weeks Using a Matching-Adjusted Indirect Comparison. Rheumatol Ther. 2024 Jun;11(3):817-828. doi: 10.1007/s40744-024-00652-7. Epub 2024 Mar 6. PMID 38446397